Study Title Duration of Dual Anti-Platelet Therapy in

**Acute Coronary Syndrome** 

The DUAL-ACS Trial

Document Title UK Consent Form

Document Version and Date Version 4.0 29 July 2020

NCT Number NCT03252249



DUAL-ACS Trial CF V4.0 29 July 2020 IRAS Project ID: 214831

## **CONSENT FORM - The DUAL-ACS Trial**

| Partic | ipant Number: | | | | |
|---|---|---|---|---|---|
| 1. | <ol> <li>I confirm that I have read and understand the participant information sheet (V4.0 22 March 2021) and the data protection information sheet (V3.0 24 July 2020) for this study and have had a chance to consider the information and ask questions.</li> </ol> | | | | |
| 2. | I understand that taking part is voluntary and that I am free to leave at any time without giving any reason and without my medical care and/or legal rights being affected. | | | | |
| 3. | I understand that individuals from the Sponsor, from the NHS or regulatory authorities may look at the sections of my medical records relevant to me taking part in this research and data collected during the study. I give them permission to look at my data and/or medical records. | | | | |
| 4. | I give permission for my personal information (including name, address, date of birth and consent form) to be passed to the University of Edinburgh and/or Edinburgh Clinical Trials Unit so the study can be administered. | | | | |
| 5. | I understand that information about my health which is held and managed by central NHS bodies and NHS Health Boards will be looked at during and after the study. To do this, I understand that my information will be shared with those bodies. | | | | |
| 6. | I give permission for my National Health Service (NHS) Number or Community Health Index (CHI) number to be collected and passed to the University of Edinburgh and/or Edinburgh Clinical Trials Unit. | | | | |
| 7. | I agree to you telling my GP I'm taking part in the study. | | | | |
| 8. | I agree to future ethically approved studies using my data (optional – please initial either the Yes or No box). | | | | Yes No |
| 9. | I agree to take part in this study | | | | |
| | Name of P | articipant | Signature | Date | |
| | | • | J | = -: <b>···</b> | |
| | Name of Person | taking consent | Signature | Date | |

1x original – into Site File; 1x copy – to Participant; 1x copy – into medical record